CLINICAL TRIAL: NCT05330000
Title: Comparative Study on Tolerance and Pharmacokinetics of Voriconazole for Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: QL-YZ1-004-001
Record Dates: First submitted 2022-02-21; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Healthy Adults
Keywords: Voriconazole; Pharmacokinetics; Tolerance
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Intervention Model Description: A total of 48 healthy adult subjects were enrolled; Intravenous drip Voriconazole (T) for injection or reference preparation vfend ® （R）in fasting state per cycle； After a 7-day cleaning period, the second cycle of cross administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voriconazole (R) (Active Comparator)
  Interventions: Drug: 4 mg/kg Voriconazole; Drug: 6 mg/kg Voriconazole
- Voriconazole (T) (Experimental)
  Interventions: Drug: 4 mg/kg Voriconazole; Drug: 6 mg/kg Voriconazole

INTERVENTIONS:
Drug: 4 mg/kg Voriconazole — Low dose group: 24 healthy adult subjects are planned to be enrolled. Intravenous drip Voriconazole for injection in fasting state per cycle. The dosage was 4 mg / kg for 80 min.
Drug: 6 mg/kg Voriconazole — High dose group: 24 healthy adult subjects are planned to be enrolled. Intravenous drip Voriconazole for injection in fasting state per cycle. The dosage was 6 mg / kg for 120 min.

SUMMARY:
A single intravenous drip of voriconazole for injection developed by Qilu Pharmaceutical (Hainan) Co., Ltd. and the original product "vfend" was given to healthy subjects ， The pharmacokinetic differences and tolerance of the two preparations were evaluated at the doses of 4mg / kg and 6mg / kg.

DETAILED DESCRIPTION:
Low dose group: 24 healthy adult subjects are planned to be enrolled. Intravenous drip Voriconazole (T) for injection or reference preparation vfend ® (R) in fasting state per cycle. The dosage was 4 mg / kg for 80 min;After a 7-day cleaning period, the second cycle of cross administration.

High dose group: 24 healthy adult subjects are planned to be enrolled. Intravenous drip Voriconazole (T) for injection or reference preparation vfend ® (R) in fasting state per cycle. The dosage was 6 mg / kg for 120 min;After a 7-day cleaning period, the second cycle of cross administration.

ELIGIBILITY:
Inclusion Criteria:

* 1) Chinese healthy adult male and female subjects aged 18-45 years (including 18 and 45 years);
* 2) The weight of male subjects shall not be less than 50kg and that of female subjects shall not be less than 45kg. Body mass index (BMI)= body weight (kg) / height 2 (M2), body mass index in the range of 19 ~ 28 kg / m2 (including critical value);
* 3) Good health: no heart, liver, kidney, digestive tract, endocrine, blood system, respiratory system and nervous systemMedical history of general, mental and metabolic abnormalities, physical examination, ECG, vital signs evaluation and experiment. The laboratory examination and other relevant examinations are normal or abnormal, have no clinical significance, and are judged as qualified by the research doctor (creatinine is not higher than the upper limit of normal value and / or liver function (alanine aminotransferase, aspartate aminotransferase, bilirubin) Not more than 1.5 × ULN）；
* 4) The subjects had no family planning and were able to take effective contraceptive measures within 6 months from the screening of the trial to the end of the study;
* 5) Voluntarily sign the informed consent form before the test, and fully understand the test content, process and possible adverse reactions Solution;
* 6) Be able to complete the research according to the requirements of the test scheme.

Exclusion Criteria:

* 1) Persons with specific allergic history (asthma, urticaria, eczema, etc.), or allergic constitution (such as for two or more drugsAllergic to food such as milk or pollen), or known allergic to this drug or similar components.
* 2) The screening results of infectious diseases (HIV antibody, hepatitis B surface antigen, hepatitis C antibody and syphilis antibody) were positive.
* 3) Female subjects in the screening period or clinical trials are in lactation or pregnancy test results are positive, or screening Whether there is protective behavior in the first 2 weeks.
* 4) Urine drug screening results were positive.
* 5) Those who have a history of drug abuse in the past five years or have used drugs in the first three months of screening.
* 6) Regular drinkers within 6 months before screening (regular drinkers are defined as drinking more than 2 units per day, or Drinking more than 14 units of alcohol a week; 1 unit = 360 ml of beer or 45 ml of 40% alcohol Wine or 150 ml wine).
* 7) Those who smoked more than 5 cigarettes a day three months before screening.
* 8) Blood donation or massive blood loss (> 400 ml, except physiological blood loss in women) within three months before screening.
* 9) Those who have a history of hospitalization or surgery within three months before screening.
* 10) Those who took clinical trial drugs within three months before screening.
* 11) Any prescription drug was taken within 14 days before taking the study drug.
* 12) Took any over-the-counter drugs or herbal products within 48 hours before taking the study drug.
* 13) Ingestion of grapefruit fruit or products containing grapefruit ingredients within 72 hours before taking the study drug.
* 14) Those who ingested beverages or foods rich in caffeine or xanthine (such as coffee, strong tea, chocolate, coke, etc.) within 48 hours before taking the study medication, or took any alcoholic products or had positive alcohol breath test results.
* 15) Any drugs that inhibit or induce the metabolism of drugs in the liver within 30 days before screening (such as inducers barbiturates, carbamazepine, phenytoin, glucocorticoids, Omeprazole; inhibitors SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines, etc.).
* 16) Those who have special requirements for diet and cannot follow the unified diet (such as intolerable to standard food, etc.).
* 17) Have a history of needle syncope, blood syncope or known severe bleeding factors that can affect venous blood collection.
* 18) Those who have difficulty in intravenous drip administration.
* 19) Acute disease occurred during the pre study screening phase or before study medication.
* 20) According to the judgment of the researcher, it is not suitable to participate in this experiment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
AUC0-t | ± 1 minute within 4 hours. ± 3 minutes for 4-12 hours. ± 5 minutes for more than 12 hours.
  17 tubes (3ml / tube) of venous blood were collected in the low dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.33h (80min, at the end of administration), 1.42h (85min), 1.5h, 1.75h, 2.0h, 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  18 tubes (3ml / tube) of venous blood were collected in the high-dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.5h, 1.75h, 2.0h (at the end of administration), 2.08h (125min), 2.17h (130min), 2.33h (140min), 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  The plasma concentration of voriconazole was determined by LC-MS / MS. Winnonlin ® 6.4 calculate the pharmacokinetic parameters.
AUC0-∞ | ± 1 minute within 4 hours. ± 3 minutes for 4-12 hours. ± 5 minutes for more than 12 hours.
  17 tubes (3ml / tube) of venous blood were collected in the low dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.33h (80min, at the end of administration), 1.42h (85min), 1.5h, 1.75h, 2.0h, 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  18 tubes (3ml / tube) of venous blood were collected in the high-dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.5h, 1.75h, 2.0h (at the end of administration), 2.08h (125min), 2.17h (130min), 2.33h (140min), 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  The plasma concentration of voriconazole was determined by LC-MS / MS. Winnonlin ® 6.4 calculate the pharmacokinetic parameters.
Cmax | ± 1 minute within 4 hours. ± 3 minutes for 4-12 hours. ± 5 minutes for more than 12 hours.
  17 tubes (3ml / tube) of venous blood were collected in the low dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.33h (80min, at the end of administration), 1.42h (85min), 1.5h, 1.75h, 2.0h, 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  18 tubes (3ml / tube) of venous blood were collected in the high-dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.5h, 1.75h, 2.0h (at the end of administration), 2.08h (125min), 2.17h (130min), 2.33h (140min), 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  The plasma concentration of voriconazole was determined by LC-MS / MS. Winnonlin ® 6.4 calculate the pharmacokinetic parameters.
Tmax | ± 1 minute within 4 hours. ± 3 minutes for 4-12 hours. ± 5 minutes for more than 12 hours.
  17 tubes (3ml / tube) of venous blood were collected in the low dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.33h (80min, at the end of administration), 1.42h (85min), 1.5h, 1.75h, 2.0h, 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  18 tubes (3ml / tube) of venous blood were collected in the high-dose group. 3ml of venous blood was collected from the contralateral upper arm at 0:00 (within 1 hour before administration) and 0.50h, 1.0h, 1.5h, 1.75h, 2.0h (at the end of administration), 2.08h (125min), 2.17h (130min), 2.33h (140min), 2.5h, 3.0h, 4.0h, 6.0h, 8.0h, 12.0h, 24.0h, 36.0h and 48.0h after administration.
  The plasma concentration of voriconazole was determined by LC-MS / MS. Winnonlin ® 6.4 calculate the pharmacokinetic parameters.

SECONDARY OUTCOMES:
Adverse event | Up to two years.
  All adverse events (clinical symptoms, signs or diseases) occurring during the test (including cleaning period) shall be recorded in the source file. The signs and symptoms, occurrence date and time, duration, end date and time, measures taken and follow-up of adverse events shall also be recorded.
female pregnancy test | Day 16 after administration.
  Urine pregnancy examination was performed during the screening period. Blood pregnancy tests were performed at the end of the study or early termination of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Doctor, Principal Investigator — National Medical Products Administration
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shanndong, China

REFERENCES:
- [Derived] Li X, Wang C, Shi P, Liu Y, Tao Y, Lin P, Li T, Hu H, Sun F, Liu S, Fu Y, Cao Y. Pharmacokinetics and safety of two Voriconazole formulations after intravenous infusion in two doses in healthy Chinese subjects. BMC Pharmacol Toxicol. 2023 Mar 3;24(1):14. doi: 10.1186/s40360-023-00652-3. PMID 36869387